CLINICAL TRIAL: NCT04128878
Title: Improvement in Endothelial Dysfunction After Initiation of Anti-arrhythmic Therapy in Atrial Fibrillation Patients
Status: Completed | Type: Observational
Sponsor: Samir Saba (Other)
Responsible Party: Sponsor-Investigator, Samir Saba, Chief, Division of Cardiology, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Other Study IDs: STUDY18090003
Record Dates: First submitted 2019-10-14; First posted 2019-10-16 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Sotalol; dofetilide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Atrial Fibrillation Cohort: Adult patients with known or new diagnosis of either paroxysmal or persistent atrial fibrillation seen at the electrophysiology outpatient clinic and admitted to the electrophysiology service for initiation of anti-arrhythmic medications (dofetilide or sotalol).
  Interventions: Drug: Sotalol; Drug: Dofetilide

INTERVENTIONS:
Drug: Sotalol — The primary goal of the study will be to evaluate the change in endothelial function seen after initiating anti-arrhythmic medical therapy. Testing will be performed at baseline prior to the 1st dose of anti-arrhythmic therapy and again 1-3 months later at outpatient follow-up visit. We will record the resting flow (RF), biological zero (BZ) and peak flow (PF) as perfusion units (PU). Specifically, we will assess arterial stiffness and vasodilation in response to acetylcholine iontophoresis, nitroprusside iontophoresis, local thermal hyperemia and reactive hyperemia. Laser speckle contrast imaging will be employed to evaluate the microvasculature. SphygmoCor (arterial tonometry) will be used to assess macrovasculature.
Drug: Dofetilide — Same as described above with sotalol.

SUMMARY:
This is a prospective, observational study that will examine endothelial dysfunction in atrial fibrillation before and after treatment with anti-arrhythmic agents and the extent to which baseline endothelial dysfunction improves after treatment.

DETAILED DESCRIPTION:
This will be a prospective, observational study and roughly 60 patients will be recruited based on strict inclusion/exclusion criteria. Goal population includes adult patients with a diagnosis of paroxysmal or persistent atrial fibrillation seen in the electrophysiology clinic and admitted to the UPMC Presbyterian electrophysiology service for initiation of anti-arrhythmic medications.

The primary goal of the study will be to evaluate the degree of endothelial function recovery seen after initiating anti-arrhythmic medical therapy. We will assess genetic markers, arterial stiffness and vasodilation in response to acetylcholine iontophoresis, nitroprusside iontophoresis, local thermal hyperemia and reactive hyperemia. Laser speckle contrast imaging will be employed to evaluate the microvasculature. SphygmoCor (arterial tonometry) will be used to assess macrovasculature. Testing will be performed at baseline prior to the 1st dose of anti- arrhythmic therapy and repeated again 1-3 months later at outpatient follow-up visit. Additionally, follow-up phone calls or office visits will take place at 6 and 12 months after the initial data collection visit to document recurrence rate of atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-75 years of age) with paroxysmal or persistent atrial fibrillation
* Patients who recovered from prior tachycardia induced cardiomyopathy will be allowed to enroll in the study.

Exclusion Criteria:

Exclusion criteria will include:

* age >75 years
* history of cardiomyopathy
* history of severe cardiac valvular disease
* history of coronary artery disease
* pulmonary artery hypertension
* congenital heart disease
* history of stroke
* chronic hypoxia
* recent worsening or flare up of obstructive or restrictive lung disease
* liver cirrhosis
* stage three or worse chronic kidney disease
* any major trauma or surgery within the preceding 3 months
* uncontrolled hyperthyroidism
* uncontrolled hypertension
* uncontrolled diabetes mellitus
* active malignancy
* poorly controlled connective tissue disease
* any acute or chronic inflammatory or infectious disease
* Patients who are already on class I or class III antiarrhythmic agents will be excluded from the study
* Patients on non-dihydropyridine calcium channel blockers and beta blockers will not be excluded from the study, as these agents are not considered anti-arrhythmics and are not hypothesized to affect endothelial function.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with known or new diagnosis of either paroxysmal or persistent atrial fibrillation seen at the electrophysiology outpatient clinic and admitted to the electrophysiology service for initiation of anti-arrhythmic medications.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Change in microvascular endothelium dependent dilation following anti-arrhythmic therapy as measured in perfusion units | 1 year
  Change in microvascular endothelium dependent dilation (in response to acetylcholine) assessed with laser speckle contrast imaging after initiating antiarrhythmic medical therapy.

SECONDARY OUTCOMES:
Correlation between microvascular endothelial dysfunction measured at baseline and atrial fibrillation recurrence. | 1 year
Correlation between microvascular endothelial function improvement with antiarrhythmic medications and atrial fibrillation recurrence. | 1 year
Correlation between microvascular endothelial function and atrial fibrillation severity represented by left atrial size and type of Afib (paroxysmal vs persistent). | 1 year
Change in other vasodilation dysfunction indices measured after initiating antiarrhythmic medical therapy. | 1 year
Correlation between vasodilation dysfunction indices measured at baseline and atrial fibrillation recurrence. | 1 year
Whether missense mutation in Cyb5R3 T117S can predict atrial fibrillation recurrence. | 1 year
Whether missense mutation in Cyb5R3 T117S is correlated with atrial fibrillation severity. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Samir Saba, MD, Principal Investigator — Chief, Division of Cardiology, University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center - Presbyterian University Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No